CLINICAL TRIAL: NCT04248712
Title: A Phase II, Randomized, Placebo-controlled Study Evaluating the Efficacy of Antihistamines in the Treatment of Eosinophilic Esophagitis (the ATEE Study)
Brief Title: Antihistamines in Eosinophilic Esophagitis
Acronym: ATEE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low enrollment
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Dawn Francis, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19-005510
Record Dates: First submitted 2020-01-28; First posted 2020-01-30 (Actual); Results first posted 2022-12-20 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-11

CONDITIONS: Eosinophilic Esophagitis
MeSH Terms: conditions — Eosinophilic Esophagitis | interventions — Famotidine; Loratadine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Participants receive Famotidine 40 mg tab twice daily by mouth and Loratadine 10 mg tab once daily by mouth for 12 weeks.
  Interventions: Drug: Famotidine; Drug: Loratadine
- Placebo Group (Placebo Comparator): Participants receive Famotidine placebo tablet matching Famotidine orally twice daily for 12 weeks, and Loratadine placebo tablet matching Loratadine orally daily for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Famotidine — 40 mg tab twice daily by mouth for 12 week duration
  Arms: Treatment Group
Drug: Loratadine — 10 mg tab once daily by mouth for 12 week duration
  Arms: Treatment Group
Drug: Placebo — Contains no active ingredient
  Arms: Placebo Group

SUMMARY:
Researchers are assessing the safety and effectiveness of antihistamines in the treatment of eosinophilic esophagitis.

DETAILED DESCRIPTION:
The purpose of this research is to determine if antihistamines are safe and effective for the treatment of eosinophilic esophagitis. Antihistamines are frequently used for the treatment of gastroesophageal reflux disease and allergic disorders, and we hypothesize they will be effective in the treatment of eosinophilic esophagitis as well. The two antihistamines used in this study are loratadine and famotidine.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18, male and female.
* Patients who carry the diagnosis of Eosinophilic Esophagitis (EoE) based on esophageal biopsies obtained within 6 months prior to enrollment (>15 eosinophils per hpf on at least 2 esophageal levels)
* Subjects must be able to give appropriate informed consent

Exclusion Criteria:

* Not willing or able to sign consent.
* Patients who have used topical or systemic corticosteroid therapy for any reason in the previous 6 weeks.
* Patients who have been treated with acid-suppressing medications (PPI or H2 receptor antagonists) in the previous 6 weeks.
* Patients on immunosuppressive or immunomodulating medications in the previous 6 weeks.
* Patients with known allergies or hypersensitivity to anti-histamines.
* Patients who have contraindications to the procurement of esophageal biopsies including patients who have known bleeding disorders, a history of bleeding diathesis, or who are currently using warfarin or clopidogrel.
* Patients who have a contraindication to the performance of an esophagogastroduodenoscopy (EGD) including previous cardiopulmonary arrest during an endoscopic procedure.
* Patients who are pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-07-10 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Francis, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Group: Participants received Famotidine 40 mg tab twice daily by mouth and Loratadine 10 mg tab once daily by mouth for 12 weeks.
  Famotidine: 40 mg tab twice daily by mouth for 12 week duration
  Loratadine: 10 mg tab once daily by mouth for 12 week duration
- Placebo Group: Participants received Famotidine placebo tablet matching Famotidine orally twice daily for 12 weeks, and Loratadine placebo tablet matching Loratadine orally daily for 12 weeks.
  Placebo: Contains no active ingredient
Period: Overall Study
Arm/Group | Treatment Group | Placebo Group
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Terminated study due to low enrollment. No subjects enrolled in the Placebo group
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Group | Placebo Group | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Description: Number of adverse events reported
Time Frame: 12 weeks
Population: Terminated study due to low enrollment. Data collection & analysis of Treatment group only. No subjects enrolled in the Placebo group
Measure: Number; unit: adverse events
Arm/Group | Treatment Group | Placebo Group
Number analyzed (Participants) | 1 | 0
adverse events | 0 |

2. Primary Outcome: Change in Maximum Eosinophil Count
Description: Calculated by maximum eosinophils per esophagogastroduodenoscopy (EGD) high-power field (eos/hpf) after therapy with antihistamines. As measured by the percentage of change in maximum eosinophil count from baseline to 12 weeks.
Time Frame: 12 weeks
Population: Terminated study due to low enrollment. No subjects enrolled in the Placebo group
Measure: Number; unit: percentage change
Arm/Group | Treatment Group | Placebo Group
Number analyzed (Participants) | 1 | 0
percentage change | 0 |

3. Secondary Outcome: Change in Symptoms of Eosinophilic Esophagitis, as Measured by Dysphagia Symptom Questionnaire
Description: Measured by the self-reported Dysphagia Symptom Questionnaire (DSQ). The DSQ ranges from 0 to 10, with a lower score indicating less symptoms and a higher score indicating more symptoms.
Time Frame: 12 weeks
Population: Terminated study due to low enrollment. Data was not collected nor analyzed. No subjects enrolled in the Placebo group
Arm/Group | Treatment Group | Placebo Group
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change in Endoscopic Response, as Measured by the Endoscopic Reference Score
Description: Percentage of subjects with endoscopic response as measured by the Eosinophilic Esophagitis (EoE) Endoscopic Reference Score (EREFS). The score ranges from 0 to 10, with a higher score indicating worse endoscopic findings of eosinophilic esophagitis.
Time Frame: 12 weeks
Population: Terminated study due to low enrollment. Data was not collected nor analyzed. No subjects enrolled in the Placebo group
Arm/Group | Treatment Group | Placebo Group
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change in Histologic Response
Description: Percentage of subjects with histologic response of ≤15 eos/hpf on biopsy at the lower and mid esophagus
Time Frame: 12 weeks
Population: Terminated study due to low enrollment. Data was not collected nor analyzed. No subjects enrolled in the Placebo group
Arm/Group | Treatment Group | Placebo Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from baseline to end of study, approximately 12 weeks
Description: Terminated study due to low enrollment. No subjects enrolled in the Placebo group
Arm/Group | Treatment Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0

LIMITATIONS AND CAVEATS:
Terminated study due to low enrollment. No subjects enrolled in the Placebo group

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-22): https://cdn.clinicaltrials.gov/large-docs/12/NCT04248712/Prot_SAP_001.pdf